CLINICAL TRIAL: NCT00571272
Title: Longitudinal Study of Genetic Causes of Intrahepatic Cholestasis (LOGIC)
Acronym: LOGIC
Status: Suspended | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: LOGIC Study - ChiLDReN Network; U01DK103149 (NIH); U01DK103140 (NIH); U01DK103135 (NIH); U01DK084575 (NIH); U01DK084538 (NIH); U01DK084536 (NIH); U01DK062503 (NIH); U01DK062500 (NIH); U01DK062497 (NIH); U01DK062481 (NIH); U01DK062470 (NIH); U01DK062466 (NIH); U01DK062456 (NIH); U01DK062453 (NIH); U01DK062452 (NIH); U01DK062445 (NIH); U01DK062436 (NIH); U24DK062456 (NIH)
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Liver Diseases; Alagille Syndrome; Alpha 1-Antitrypsin Deficiency
Keywords: Cholestatic Liver Disease; Cholestasis; Childhood Diseases; Genetic Diseases; Bile Acid Synthesis and Metabolism Defects; Progressive Familial Intrahepatic Cholestasis
MeSH Terms: conditions — Liver Diseases; Alagille Syndrome; alpha 1-Antitrypsin Deficiency; Cholestasis; Genetic Diseases, Inborn; Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (4):
- 1: Infants less than 6 months old with a cholestatic liver disease who were initially enrolled into the Childhood Liver Disease Research and Education Network (ChiLDREN) Prospective Biliary Atresia Epidemiology study (PROBE study; P003)
- 2: Participants with a cholestatic liver disease who are between birth and 25 years old who were NOT initially enrolled into the Childhood Liver Disease Research and Education Network (ChiLDREN) Prospective Biliary Atresia Epidemiology study (PROBE study; P003)
- 3: Post-liver transplant participants with a cholestatic liver disease who are between 1 day and 25 years old. Affected parents of patients enrolled in the study are eligible for enrollment if they are 25 years old or less
- 5: Affected siblings (without evidence of liver disease) of Alpha-1 Antitrypsin Deficiency participants who are enrolled in LOGIC.

SUMMARY:
Cholestasis is a condition in which bile is not properly transported from the liver to the small intestine. Cholestasis can be caused by an array of childhood diseases, including the genetic diseases Alagille syndrome (ALGS), alpha-1 antitrypsin (a-1AT) deficiency, bile acid synthesis and metabolism defects, and progressive familial intrahepatic cholestasis (PFIC) or benign recurrent intrahepatic cholestasis(BRIC). This study will investigate the natural history and progression of the four previously mentioned cholestatic liver diseases to provide a better understanding of the causes and effects of the diseases.

DETAILED DESCRIPTION:
Cholestasis is a rare condition that involves a reduction or obstruction of bile flow from the liver to the small intestine. When bile flow is hindered, a waste product pigment called bilirubin can escape into the bloodstream and build up to harmful levels. This may lead to the easily recognizable cholestatic symptoms of jaundice, itching, and impaired growth and eventually to more serious health problems. Four rare genetic liver disorders- ALGS, a-1AT, bile acid synthesis and metabolism defects, and PFIC-account for about 20% to 30% of all infant cases of cholestasis. These four disorders compose a group of related diseases that can cause significant growth problems during childhood, serious liver problems, the need for liver transplantation, and potentially death. More research on these rare liver diseases is necessary to develop a scientific basis for improvement in diagnostic techniques and treatments. Current diagnostic procedures are complex, and the development of simpler diagnostic tests would facilitate early diagnosis and treatment. This study will investigate the natural history and progression of the four previously mentioned cholestatic liver diseases to provide a better understanding of the causes and effects of the diseases.

Participants who have been previously enrolled into this study will be followed for 20 years, until transplanted, or death. Study visits will involve review of clinical information, family history, and any clinically indicated treatments and their outcomes; a physical exam; laboratory tests; and radiologic and imaging evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Children and young adults diagnosed with one of the four cholestatic diseases from birth through 25 years old.
2. Siblings of participants with alpha-1-antitrypsin deficiency, who are affected with alpha-1-antitrypsin deficiency, but have no evidence of liver disease.
3. Both sexes, all races and ethnic groups.
4. Participant meets the enrollment criteria for one of the four cholestatic liver diseases.
5. Patient and/or parent/legal guardian have the ability to provide written informed consent for enrollment.

Exclusion Criteria:

1. Inability to comply with the longitudinal follow-up described in the protocol.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will consist of 400 participants with Alagille syndrome, 400 with alpha-1 trypsin deficieny (of which up to 25 may be siblings of participants), 300 with PFIC (or BRIC), and 50 with bile acid synthesis defects.
Sampling Method: Non-Probability Sample
Enrollment: 1675 (Estimated)
Dates: Start 2007-11-30 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Demonstration of disease progression for each of the four cholestatic liver diseases of the study, including liver transplantation, death, growth failure, worsening liver function, and developmental complications of portal high blood pressure | Measured at baseline and annually through year 10

SECONDARY OUTCOMES:
Jaundice (total serum bilirubin of greater than 2.0 mg/dl) | Measured at baseline and annually through year 10
Listing for liver transplantation | Measured at baseline and annually through year 10
Calculated Pediatric End-Stage Liver Disease (PELD) score for participants less than 12 years of age or Model for End-Stage Liver Disease (MELD) score for participants 12 years of age or older | Measured at baseline and annually through year 10
Health related quality of life | Measured at baseline and annually through year 10
Growth (length and weight Z-score) | Measured at baseline and annually through year 10
Bone mineral density (lumbar and spine total body) | Measured at baseline in ALGS and PFIC/BRIC subjects
Presence of hearing loss (ALGS and PFIC) | Measured at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Loomes, MD, Study Chair — Children's Hospital of Philadelphia; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John Magee, MD, Principal Investigator — University of Michigan; Lisa Henn, PhD, Principal Investigator — Arbor Research Collaborative for Health; Katrina Loh, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (17):
- United States (16):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California at San Francisco (UCSF), San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - St. Louis University - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine/St. Louis Children's Hospital, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Cincinnati's Children's Memorial Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor School of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data will be transferred to NIDDK at the end of the study.

REFERENCES:
- [Derived] Teckman J, Rosenthal P, Ignacio RV, Spino C, Bass LM, Horslen S, Wang K, Magee JC, Karpen S, Asai A, Molleston JP, Squires RH, Kamath BM, Guthery SL, Loomes KM, Shneider BL, Sokol RJ; ChiLDReN (Childhood Liver Disease Research Network). Neonatal cholestasis in children with Alpha-1-AT deficiency is a risk for earlier severe liver disease with male predominance. Hepatol Commun. 2023 Dec 7;7(12):e0345. doi: 10.1097/HC9.0000000000000345. eCollection 2023 Dec 1. PMID 38055647
- [Derived] Leung DH, Sorensen LG, Ye W, Hawthorne K, Ng VL, Loomes KM, Fredericks EM, Alonso EM, Heubi JE, Horslen SP, Karpen SJ, Molleston JP, Rosenthal P, Sokol RJ, Squires RH, Wang KS, Kamath BM, Magee JC; Childhood Liver Disease Research Network (ChiLDReN). Neurodevelopmental Outcomes in Children With Inherited Liver Disease and Native Liver. J Pediatr Gastroenterol Nutr. 2022 Jan 1;74(1):96-103. doi: 10.1097/MPG.0000000000003337. PMID 34694263
- [Derived] Teckman JH, Rosenthal P, Abel R, Bass LM, Michail S, Murray KF, Rudnick DA, Thomas DW, Spino C, Arnon R, Hertel PM, Heubi J, Kamath BM, Karnsakul W, Loomes KM, Magee JC, Molleston JP, Romero R, Shneider BL, Sherker AH, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Baseline Analysis of a Young alpha-1-Antitrypsin Deficiency Liver Disease Cohort Reveals Frequent Portal Hypertension. J Pediatr Gastroenterol Nutr. 2015 Jul;61(1):94-101. doi: 10.1097/MPG.0000000000000753. PMID 25651489
- See also: Childhood Liver Disease Research Network (ChiLDReN) website — http://www.childrennetwork.org